CLINICAL TRIAL: NCT04066049
Title: EMT en Español: Comprehensive Early Intervention to Support School Readiness Skills for Spanish-speaking Toddlers With Language Delays
Brief Title: EMT en Español for Spanish-speaking Toddlers With Language Delays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ann Kaiser, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R324A190177
Record Dates: First submitted 2019-08-07; First posted 2019-08-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Language Development Disorders
Keywords: Spanish-speaking; caregiver-implemented intervention; bilingual
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: Participants in the Treatment group will receive a hybrid therapist-implemented and caregiver-implemented intervention and be compared to a BAU control group. Caregivers and children will be assessed at baseline, after the intervention, 6 months after intervention, and 12 months after intervention.
Who Masked: Outcomes Assessor
Masking Description: Standardized and observational measures will be conducted by independent observers and assessors (master's level bilingual speech-language pathologists) who are blind to the experimental conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Participants in the Treatment group will receive a hybrid therapist-implemented and caregiver-implemented intervention be compared to a BAU control group. Caregivers and children will be assessed at baseline, after the intervention, 6 months after intervention, and 12 months after intervention, and will receive a $50 gift card for participating in each assessment time point, $75 for completing all four assessments, and books and play/activity materials with target word lists in Spanish.
  Interventions: Behavioral: EMT en Español
- Control (No Intervention): Participants in the BAU group will be offered 10 caregiver support sessions after completing the 12-month follow-up. These home-based sessions will emphasize shared book reading, modeling vocabulary for school readiness in play and routines, and include general information for families about options for public school language related services. Each session will last about 30 minutes and be conducted by a trained staff member. Caregivers and children will be assessed at baseline, after the intervention, 6 months after intervention, and 12 months after intervention, and will receive a $50 gift card for participating in each assessment time point, $75 for completing all four assessments, and books and play/activity materials with target word lists in Spanish.

INTERVENTIONS:
Behavioral: EMT en Español — EMT en Español utilizes intervention strategies adapted from Enhanced Milieu Teaching (Kaiser & Hampton, 2016), an evidence-based naturalistic communication intervention, to promote home language and improve children's language use across the day in home routines, play, and book sharing in individual sessions with a therapist and in caregiver training sessions.
  Arms: Treatment

SUMMARY:
The goal of the study is to conduct an initial efficacy study of a promising therapist and caregiver-implemented communication intervention to improve language and school readiness skills in low-income Spanish-speaking children with receptive and expressive language delays (ages 30 to 36 months). The proposed randomized trial compares the effects of a caregiver plus therapist implemented EMT en Español intervention to a community based "business as usual" control group at four time points (pre- intervention, post-intervention, 6 month follow-up, 12 month follow-up) in a sample of 84 low-income, Spanish-speaking families and their toddlers with receptive and expressive language delays.

DETAILED DESCRIPTION:
The goal of the study is to conduct an initial efficacy study of a promising therapist and caregiver-implemented communication intervention to improve language and school readiness skills in low-income Spanish-speaking children with receptive and expressive language delays (ages 30 to 36 months). This randomized trial compares the effects of a caregiver plus therapist implemented EMT en Español intervention to a community based "business as usual" control group at four time points (pre- intervention, post-intervention, 6 month follow-up, 12 month follow-up) in a sample of 84 low-income, Spanish-speaking families and their toddlers with receptive and expressive language delays.

The target population of children for this study is multiply at-risk for persistent language delays and later language-related academic difficulties. First, before age three, the identified children have significant delays in both receptive and expressive language abilities. Significant delays in both domains of language by 30 months of age places children at-risk for persistent language impairment at school entry and beyond. Second, these children's families are low-income ethnic minorities residing in the U.S. As such, these families and children are more likely to live in segregated communities with limited neighborhood resources, poorer quality schools, and less access to quality health care. Finally, these children's caregivers are Spanish-speaking immigrants who are likely to face discrimination based on their own language use and to face cultural and linguistic barriers in accessing needed services for their children. We note that the population for this study differs from children who are considered at-risk because they are from low-income ethnic minority families. The target population for this project is young children who already evidence significant delays in both language understanding and production in addition to coming from low-income families. This is a population for whom there are no current evidence-based interventions and for whom early, effective language intervention is essential to their later academic learning. The intervention, EMT en Español, utilizes intervention strategies adapted from Enhanced Milieu Teaching, an evidence-based naturalistic communication intervention, to promote home language and improve children's language useacross the day in home routines, play, and book sharing in individual sessions with a therapist and in caregiver training sessions. The current study builds on two preliminary studies of EMT in Español and evidence from an RCT of EMT with English-speaking toddlers with receptive and expressive language delays. The caregiver training component of the intervention utilizes an evidence-based caregiver instruction and coaching protocol to deliver the EMT en Español intervention in families' homes in Spanish.

A randomized clinical trial (RCT) design is proposed to compare the effects of EMT in Español to a community business as usual (BAU) control group. The immediate and long-term effects of the intervention on children's language development and on their caregivers' use of naturalistic teaching strategies including linguistic input will be examined over the 18 months of the study. Note that the population of children for this study are monolingual Spanish-speakers at30 months, who may have some limited exposure to English. Children in this study will likely be dual language learners when they enter preschool. All outcomes and measures account for children's language abilities across languages.

ELIGIBILITY:
Inclusion Criteria:

* Spanish is the primary language spoken to the child by caregivers as measured by the Home Language Scale
* The child demonstrates expressive and receptive language delays (at least 1.5 standard deviations below the mean n each domain as measured on the Preschool Language Scale- 5th edition Spanish)
* The child demonstrates cognitive skills within 1 standard deviation of the mean as measured by the Leiter-R
* The child is between 30-36 months old
* The child does not have any other disabilities (e.g. ASD, Down syndrome, cerebral palsy, blindness, deafness)
* There is one consistent caregiver willing to participate in training and assessments
* The family meets criteria for low-income status (i.e., income is up to 2 times federal poverty level for a family of that size)

Exclusion Criteria:

* Spanish is not primary language spoken to the child by caregiver as measured by the Home Language Scale
* The child does not demonstrate expressive and receptive language delays (at least 1.5 stand deviations below the mean n each domain as measured on the Preschool Language Scale- 5th edition Spanish)
* The child does not demonstrate cognitive skills within 1 standard deviation of the mean as measured by the Leiter-R
* The child is over 36 months old
* The child has another disability (e.g. ASD, Down syndrome, cerebral palsy, blindness, deafness)
* There is not a consistent caregiver willing to participate in training and assessments
* The family does not meet criteria for low-income status (i.e. income is more than 2 times the federal poverty level for a family of that size)

Ages: 30 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Unprompted Number of Different Conceptual Words across English and Spanish from 2 20-minute standardized play-based Language Samples with a trained assessor. | 5 months
  The non-imitated, non-prompted number of different conceptual words spoken by the child across Spanish and English taken from a combined sample of 1 20-minute play-based Language Sample administered in Spanish and 1 20-minute play-based Language Sample administered in English.
Number of language targets used across 2 20-minute standardized play-based language samples with a trained assessor. | 5 months
  The number of specific language targets in English and Spanish, including words and phrases individualized to the child based on their level of language, taken from a combined sample of 1 20-minute play-based Language Sample administered in Spanish and 1 20-minute play-based Language Sample administered in English.
Total raw score from Receptive and Expressive One-Word Picture Vocabulary Tests - Spanish Bilingual Edition (ROWPVT-SBE) | 5 months
  Minimum Total Raw Score: 0; Maximum Total Raw Score: 180; Higher scores are considered better outcomes.

OTHER OUTCOMES:
Bilingual English-Spanish Assessment (BESA) standard score (0-100) | 17 months
  The BESA is designed to be used with children who speak English, Spanish, or both.
  The BESA subtests are psychometrically sound and yield scaled and standard scores for each of the domain tests (phonology, morphosyntax, and semantics). The BESA is specifically designed to assess speech and language in English-Spanish bilingual children's two languages. The primary use of the BESA is to identify phonological and/or language impairment in bilingual and English language learner (ELL) children via a standardized protocol. The objective scores obtained on the BESA across three domains can be used in combination with clinical observations and language samples, as well as with other standardized measures, to identify children with speech and/or language impairment. Through use of a combination of BESA subtests, clinicians can document children's speech and language strengths and weaknesses.
  A higher score is considered better than a lower score.
Composite Executive Function Score | 5 months, 11 months, 17 months
  Composite executive function score taken from a Snack Delay Task and Head-Shoulders-Knees-Toes (HSKT) administered by a trained assessor, and the Behavior Rating Inventory of Executive Function Preschool (BRIEF-P) Spanish completed by the parent. The Snack Delay Task and BRIEF-P are administered at 5 months, 11 months and 17 months. The HSKT is only administered at 17 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ann P Kaiser, PhdD, Principal Investigator — Vanderbilt University; Tatiana Peredo, PhdD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT04066049/ICF_000.pdf